CLINICAL TRIAL: NCT05748015
Title: Definition of Autonomic Nervous System Involvement in Patients With Relapsing-remitting and Primary Progressive Multiple Sclerosis
Brief Title: Definition of Autonomic Nervous System Involvement in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SBLAB/SM20
Record Dates: First submitted 2023-01-26; First posted 2023-02-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: autonomic nervous system; sensory nervous system; rehabilitation; skin biopsy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relapsing-remitting multiple sclerosis (Active Comparator): Patients with relapsing-remitting multiple sclerosis will be hospitalized in Maugeri Clinical Institute of Telese Terme for a rehabilitation treatment and will perform a functional and morphological study of sensory and autonomic nervous system, evaluation of peripheral sensory and autonomic nerve fibers performed by skin biopsy.
  Interventions: Diagnostic Test: quantification of sensory and autonomic small nerve fibers by punch skin biopsy; Diagnostic Test: Cardiovascular Reflexes testing; Other: Administration of clinical scales evaluating autonomic symptoms, pain small fiber neuropathy symptoms
- primary progressive multiple sclerosis (Active Comparator): Patients with primary progressive multiple sclerosis will be hospitalized in Maugeri Clinical Institute of Telese Terme for a rehabilitation treatment and will perform a functional and morphological study of sensory and autonomic nervous system, evaluation of peripheral sensory and autonomic nerve fibers performed by skin biopsy.
  Interventions: Diagnostic Test: quantification of sensory and autonomic small nerve fibers by punch skin biopsy; Diagnostic Test: Cardiovascular Reflexes testing; Other: Administration of clinical scales evaluating autonomic symptoms, pain small fiber neuropathy symptoms

INTERVENTIONS:
Diagnostic Test: quantification of sensory and autonomic small nerve fibers by punch skin biopsy — We'll perform a punch skin biopsy of 3mm from thigh, leg and fingertip and we'll quantify peripheral sensory and autonomic nerve fibers.
Diagnostic Test: Cardiovascular Reflexes testing — Cardiovascular reflex tests including deep breathing, head-up Tilt, standing, isometric exercises, mental arithmetic and Valsalva maneuver.
Other: Administration of clinical scales evaluating autonomic symptoms, pain small fiber neuropathy symptoms — We'll characterize patients' symptoms through the administration of clinical scales such as: COMPASS 31 autonomic symptoms scale; Small Fiber Neuropathy Symptom Inventory Questionnaire (SFN-SIQ), the Pain Detect Questionnaire and the Total neuropathy score

SUMMARY:
The goal of this interventional non-pharmacological study is to evaluate the involvement of the autonomic nervous system in patients with relapsing-remitting and primary progressive multiple sclerosis.

The main questions it aims to answer are:

* Is it possible to define the characteristics of dysautonomia to improve treatment on patients with multiple sclerosis through the management of conditions such as orthostatic hypotension or thermoregulation disorders that inevitably condition the patient's life and the response to rehabilitation ?
* Does the severity of the functional alterations correlate with impairment of small somatic and autonomic cutaneous nerve fibers in patients with multiple sclerosis ?
* How much the involvement of the autonomic nervous system affects the clinical history and progression of the disease ?
* Do different clinical variants of multiple sclerosis manifest with different patterns of involvement of the sensory-autonomic nervous system ?

Participants will be hospitalized in Maugeri Clinical Institute of Telese Terme for a rehabilitation treatment. Patients will perform a sensory and autonomic functional study and a morphological analysis of cutaneous nerves through skin biopsy.

Researchers will compare results between the two groups (relapsing-remitting and primary progressive) and between patients and data from control subjects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsing-remitting and primary progressive multiple sclerosis.

Exclusion Criteria:

* other forms of multiple sclerosis,
* known other neurological disorders
* assumption of potentially neurotoxic substances or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular reflex test | At the recruitment
  Assessment of Cardiovascular reflex responses to physical challenges.
Sudomotor function test | At the recruitment
  Assessment of postganglionic sudomotor function through dynamic sweat test

SECONDARY OUTCOMES:
Quantification of peripheral autonomic nerve fibers | At the recruitment
  Quantification of sweat gland innervation (fiber length /um3) and arrector pili muscle (ff/mm).
Quantification of peripheral sensory nerve fibers | At the recruitment
  Quantification of sensory nerve fibers (Intraepidermal nerve fibers (ff/mm)).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Provitera, MD, Principal Investigator — ICS MAUGERI - IRCCS TELESE TERME
Locations (2):
- Italy (2):
  - ICS Maugeri - IRCCS of Telese Terme, Telese Terme, Benevento
  - Department of Neurosciences, Reproductive Sciences and Odontostomatology, University of Naples Federico II, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahoney CJ, Ahmed RM, Huynh W, Tu S, Rohrer JD, Bedlack RS, Hardiman O, Kiernan MC. Pathophysiology and Treatment of Non-motor Dysfunction in Amyotrophic Lateral Sclerosis. CNS Drugs. 2021 May;35(5):483-505. doi: 10.1007/s40263-021-00820-1. Epub 2021 May 15. PMID 33993457
- [Background] Gentile F, Scarlino S, Falzone YM, Lunetta C, Tremolizzo L, Quattrini A, Riva N. The Peripheral Nervous System in Amyotrophic Lateral Sclerosis: Opportunities for Translational Research. Front Neurosci. 2019 Jun 25;13:601. doi: 10.3389/fnins.2019.00601. eCollection 2019. PMID 31293369
- [Background] Weis J, Katona I, Muller-Newen G, Sommer C, Necula G, Hendrich C, Ludolph AC, Sperfeld AD. Small-fiber neuropathy in patients with ALS. Neurology. 2011 Jun 7;76(23):2024-9. doi: 10.1212/WNL.0b013e31821e553a. PMID 21646630
- [Background] Truini A, Biasiotta A, Onesti E, Di Stefano G, Ceccanti M, La Cesa S, Pepe A, Giordano C, Cruccu G, Inghilleri M. Small-fibre neuropathy related to bulbar and spinal-onset in patients with ALS. J Neurol. 2015;262(4):1014-8. doi: 10.1007/s00415-015-7672-0. Epub 2015 Feb 17. PMID 25683764
- [Background] Nolano M, Provitera V, Manganelli F, Iodice R, Caporaso G, Stancanelli A, Marinou K, Lanzillo B, Santoro L, Mora G. Non-motor involvement in amyotrophic lateral sclerosis: new insight from nerve and vessel analysis in skin biopsy. Neuropathol Appl Neurobiol. 2017 Feb;43(2):119-132. doi: 10.1111/nan.12332. Epub 2016 Jul 7. PMID 27288647
- [Background] deCarvalho M, Gromicho M, Andersen P, Grosskreutz J, Kuzma-Kozakiewicz M, Petri S, Uysal H, Pinto S. Peripheral neuropathy in ALS: phenotype association. J Neurol Neurosurg Psychiatry. 2021 Oct;92(10):1133-1134. doi: 10.1136/jnnp-2020-325164. Epub 2020 Dec 28. No abstract available. PMID 33372053
- [Background] Chio A, Mora G, Lauria G. Pain in amyotrophic lateral sclerosis. Lancet Neurol. 2017 Feb;16(2):144-157. doi: 10.1016/S1474-4422(16)30358-1. Epub 2016 Dec 8. PMID 27964824
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847